CLINICAL TRIAL: NCT07374419
Title: A Phase Ib/II Study of Atamparib in Patients With Advanced Solid Tumors
Brief Title: Atamparib in Patients With Advanced Solid Tumors
Acronym: PARP7
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nerviano Medical Sciences (Shanghai) Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRP7A-ATA-001
Record Dates: First submitted 2026-01-06; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: NSCLC Adenocarcinoma; Solid Tumor
Keywords: PRP7A-ATA-001, Atamparib; Neviano, NMS
MeSH Terms: conditions — Neuroleptic Malignant Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- monotherapy escalation (Experimental): Atamparib
  Interventions: Drug: atamparib escalation levels
- Espansion Arm a (Experimental): Atamparib
  Interventions: Drug: atamparib RP2D
- Expansion Arm b (Experimental): Atamparib
  Interventions: Drug: atamparib RP2D
- Expansion Arm c (Experimental): Atamparib
  Interventions: Drug: atamparib RP2D
- Expansion Arm d (Experimental): Atamparib
  Interventions: Drug: atamparib RP2D

INTERVENTIONS:
Drug: atamparib escalation levels — Bid, Oral, escalating at different dose levels
  Arms: monotherapy escalation
Drug: atamparib RP2D — Bid, oral, RP2D
  Arms: Espansion Arm a; Expansion Arm b; Expansion Arm c; Expansion Arm d

SUMMARY:
This is a multi-part, open-label, non-randomized phase Ib/II clinical trial designed to evaluate the safety, tolerability, pharmacokinetics, and preliminary antitumor activity of atamparib, an investigational agent, in patients with advanced or metastatic non-small cell lung cancer (NSCLC) adenocarcinoma. The study comprises dose escalation (phase Ib) and expansion (phase II).

ELIGIBILITY:
Inclusion criteria:

1. Subject must be ≥18 years of age.
2. Histologically confirmed diagnosis of unresectable advanced or metastatic NSCLC adenocarcinoma.
3. Documented KRAS mutation status at study entry.
4. Have received at least one line of standard therapy and experienced radiographic tumor progression to the last administered treatment and have failed institutional standards of care.
5. Have measurable tumor lesions
6. ECOG 0-1
7. Adequate organ functions

Exclusion criteria:

1. Non-adenocarcinoma histology of NSCLC. Patients whose tumors have a mixed histology are ineligible.
2. Wtih oncogenic driver mutation other than KRAS for which an approved therapy is available but not adequately treated.
3. Known active GI disease that would impact the absorption
4. Clinically significant cardiac disease
5. Requiring the administration of strong inhibitors or inducers of CYP3A4, P-gp or BCRP.
6. Symptomatic, or untreated CNS lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
RP2D and MTD | 28 days after the last dose
  First cycle DLTs and all other available study data
Type, incidence and severity of adverse event | until 28 days after the last dose
  Safety and tolerability profile assessed by the CTCAE v6.0

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, Dr., Principal Investigator — Shanghai East Hospital, Yuntailu 1800
Locations (1):
- Unit 3.53, 3rd Floor, No. 5, Lane 720 Cailun Road, Pilot Free Trade Zone, Shanghai, P.R.China, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided